## Testing of a Tool to Elicit Patient Preferences for CTS

Informed Consent Form

NCT03532373

March 31, 2023

## STANFORD UNIVERSITY Research Consent Form

Protocol Director: Robin Kamal, MD

Protocol Title: Testing of a tool to elicit patient preferences for CTS

IRB Use Only Approval Date: March 31, 2023 Expiration Date: March 31, 2024

FOR QUESTIONS ABOUT THE STUDY, CONTACT: Protocol Director, Robin Kamal, MD, 450 Broadway Street, Redwood City, CA 94063, 650-723-5643

**DESCRIPTION:** You are invited to participate in a research study to test a new tool to elicit patient preferences in the treatment of carpal tunnel syndrome. The tool presents various attributes of each carpal tunnel treatment, such as the cost and success rate. If you agree to participate, you may be asked to use the tool or you may not be asked to use the tool. You will be assigned to your study group by a random number generator. You will be asked to complete a survey at the end of your visit. A description of this clinical trial will available on http://clinicaltrials.gov as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search the Web site at any time.

**RISKS AND BENEFITS:** The risks associated with this study are minimal and not expected to be any greater than what you would experience in everyday life. No benefits accrue to you for participating in this study, but your responses will be used to better tailor our treatment recommendations for future patients and may help you be more confident in your decision. We cannot and do not quarantee or promise that you will receive any benefits from this study. Your decision whether or not to participate in this study will not affect your medical care.

**TIME INVOLVEMENT:** Your participation in this experiment will take approximately 5-10 minutes per visit.

**PAYMENTS:** You will not receive payment for your participation.

**PARTICIPANT'S RIGHTS:** If you have read this form and have decided to participate in this project, please understand your participation is voluntary and you have the right to withdraw your consent or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled.

**SPONSOR:** The National Institute of Health and the Orthopaedic Research and Education Foundation are providing financial support and/ or material for this study.

The results of this research study may be presented at scientific or professional meetings or published in scientific journals. However, your identity will not be disclosed. You have the right to refuse to answer particular questions.

## **CONTACT INFORMATION:**

Questions, Concerns, or Complaints: If you have any questions, concerns or complaints about this research study, its procedures, risks and benefits, or alternative courses of treatment, you should ask the Protocol Director, Robin Kamal, MD. You may contact him/her now or later at 650-723-5643. Independent Contact: If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact the Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at (650)-723-5244 or toll free at 1-866-680-2906. You can also write to the Stanford IRB, Stanford University, 1705 El Camino Real, Palo Alto, CA 94306.

The extra copy of this Research Information Sheet is for you to keep. If you agree to participate in this research, please complete the attached survey.